CLINICAL TRIAL: NCT07319663
Title: Quasi-experimental Community-Based Social Connection Intervention Program to Improve Cardiovascular and Brain Health in Older Adults Living in Rural Ecuador
Brief Title: Community-Based Social Connection Intervention Program to Improve Cardiovascular and Brain Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Especialidades Espiritu Santo (Other)
Collaborators: University of Miami (Other)
Responsible Party: Principal Investigator, Oscar H. Del Brutto, Director, the Atahualpa Project, Universidad de Especialidades Espiritu Santo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UniversidadEES
Record Dates: First submitted 2025-12-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Social Isolation in Older Adults; Loneliness; Stroke; Cognitive Decline
Keywords: Social isolation; Loneliness; Social support; Community Health Services; Rural population; Aged
MeSH Terms: conditions — Stroke; Cognitive Dysfunction; Social Isolation

STUDY DESIGN:
Intervention Model Description: This study uses a quasi-experimental, community-based longitudinal design to evaluate the impact of a social connection intervention on older adults in rural Ecuador. One community receives the intervention, while two comparable communities serve as non-randomized comparison groups. Allocation is based on pre-existing community of residence. Participants are followed for 12 months with assessments at baseline, 6 months, and 12 months. The intervention includes monthly community activities, monthly peer-support groups, and twice-monthly home-based coaching. Outcomes include social isolation, loneliness, cardiovascular health, cognition, sleep, mood, and quality of life.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention community (SCIP) (Experimental): Participants in this community receive the Social Connection Intervention Program (SCIP), which includes monthly community activities and educational talks, monthly peer-support group sessions, and twice-monthly individualized home-based coaching. The program is delivered over 12 months to reduce social isolation and loneliness and promote cardiovascular and brain health.
  Interventions: Other: Social Connection Intervention Program (SCIP): Community activities, peer-support groups, and home-based coaching to reduce social isolation and loneliness.
- control (No Intervention)

INTERVENTIONS:
Other: Social Connection Intervention Program (SCIP): Community activities, peer-support groups, and home-based coaching to reduce social isolation and loneliness. — The Social Connection Intervention Program (SCIP) is a 12-month, community-based program designed to reduce social isolation and loneliness among older adults in rural Ecuador. The intervention includes three components: (1) monthly community activities and educational talks to promote social participation and health awareness; (2) monthly peer-support group sessions facilitated by trained personnel to enhance emotional support and shared problem-solving; and (3) twice-monthly individualized home-based coaching sessions incorporating principles of Social Cognitive Theory and Cognitive Behavioral Therapy to strengthen coping skills, goal-setting, and healthy behaviors. The program is delivered in the intervention community, while comparison c
  Arms: intervention community (SCIP)

SUMMARY:
This study evaluates the effectiveness of a community-based social connection intervention program (SCIP) designed to reduce social isolation and loneliness and improve cardiovascular and brain health among older adults living in rural Ecuador. Loneliness and social isolation are recognized risk factors for poor cardiovascular outcomes, cognitive decline, depression, and reduced quality of life. However, evidence from low- and middle-income countries, particularly in rural Latin American settings, remains limited. This protocol describes a quasi-experimental, longitudinal study conducted in three rural villages that have been part of a long-standing population-based cohort.

The intervention will be implemented in one community and compared with two similar communities that will continue receiving usual community activities. SCIP consists of three components: (1) monthly community activities and educational talks designed to promote social participation; (2) monthly peer-support group sessions facilitated by trained personnel; and (3) individualized home-based coaching delivered twice per month, incorporating principles of Social Cognitive Theory and Cognitive Behavioral Therapy. The program aims to strengthen social networks, enhance coping skills, and promote healthier behaviors.

Participants aged 60 years and older will be enrolled and followed for 12 months. Assessments will occur at baseline, 6 months, and 12 months. Primary outcomes include changes in social isolation (Lubben Social Network Scale-6) and loneliness (De Jong Gierveld Scale). Secondary outcomes include cardiovascular health (Life's Essential 8), sleep quality (Pittsburgh Sleep Quality Index), cognitive performance (Montreal Cognitive Assessment), depressive symptoms (DASS-21), and quality of life (SF-36). Exploratory outcomes include incident stroke, cardiovascular events, and mortality, monitored through ongoing community surveillance.

This study will generate evidence on the feasibility and impact of a culturally adapted, community-based intervention to promote social connection and healthy aging in a resource-limited rural setting. Findings may inform scalable public health strategies for older adults in similar contexts.

DETAILED DESCRIPTION:
Loneliness and social isolation are increasingly recognized as major public health concerns, particularly among older adults. These conditions are associated with elevated risks of cardiovascular disease, cognitive decline, depression, sleep disturbances, reduced quality of life, and premature mortality. Although evidence from high-income countries supports the use of community-based interventions to enhance social connection, there is limited research in low- and middle-income countries and almost no data from rural Latin American settings. The Social Connection Intervention Program (SCIP) was developed to address this gap by adapting evidence-based strategies to the cultural, social, and resource context of rural Ecuador.

Study Design and Setting: This is a quasi-experimental, longitudinal study conducted in three rural villages in coastal Ecuador that have participated in a population-based cohort for more than 12 years. One community (Atahualpa) will receive the intervention, while two comparable communities (El Tambo and Prosperidad) will serve as comparison sites. Allocation is based on pre-existing community of residence. The study will follow participants for 12 months, with assessments at baseline, 6 months, and 12 months.

Participants: Eligible participants are adults aged 60 years or older who have lived in the community for at least one year, have no plans to relocate, and do not have disability, dementia, stroke, or major psychiatric illness. Written informed consent will be obtained from all participants. Recruitment will leverage the existing cohort infrastructure, which has historically achieved high retention rates.

Intervention: SCIP consists of three integrated components: 1. Community Activities and Educational Talks: Monthly group activities designed to promote social participation, health education, and community engagement. Activities include cultural events, group discussions, and interactive workshops; 2. Peer-Support Groups: Monthly small-group sessions facilitated by trained personnel, focusing on emotional support, shared experiences, and collective problem-solving. These sessions aim to strengthen interpersonal connections and reduce feelings of loneliness , and 3. Home-Based Coaching: Twice-monthly individualized coaching sessions delivered in participants' homes. The coaching incorporates principles of Social Cognitive Theory and Cognitive Behavioral Therapy, emphasizing goal-setting, self-efficacy, coping strategies, and behavior change to support healthier lifestyles and social engagement.

The comparison communities will continue with their usual activities and will not receive SCIP during the study period.

Outcomes: The primary outcomes are changes in social isolation and loneliness from baseline to 12 months, measured using the Lubben Social Network Scale-6 (LSNS-6) and the De Jong Gierveld Loneliness Scale. Secondary outcomes include cardiovascular health assessed through the American Heart Association's Life's Essential 8 metrics, sleep quality (Pittsburgh Sleep Quality Index), cognitive performance (Montreal Cognitive Assessment), depressive symptoms (DASS-21), and quality of life (SF-36). Exploratory outcomes include incident stroke, cardiovascular events, vascular mortality, and all-cause mortality, monitored through ongoing community surveillance.

Data Collection and Management: Data will be collected through face-to-face interviews, validated questionnaires, and standardized clinical measurements. All data will be stored in a secure, encrypted database with restricted access. Quality control procedures include periodic audits and verification of data completeness and accuracy.

Statistical Analysis: Analyses will follow an intention-to-treat approach. Mixed-effects models will be used for continuous outcomes, logistic regression or generalized estimating equations for categorical outcomes, and Cox proportional hazards models for time-to-event outcomes. Multiple imputation will be used to address missing data. Sensitivity analyses will assess the robustness of findings.

Ethics and Dissemination: The study has been approved by the Independent Review Board of Hospital-Clínica Kennedy (FWA: 00030727). Protocol amendments will be submitted to the IRB and updated in the trial registry. Results will be disseminated to the community, local health authorities, scientific conferences, and peer-reviewed journals.

This study will provide valuable evidence on the feasibility, acceptability, and effectiveness of a culturally adapted, community-based intervention to reduce loneliness and social isolation and promote cardiovascular and brain health among older adults in a resource-limited rural setting. Findings may inform scalable public health strategies for healthy aging in similar contexts.

ELIGIBILITY:
Inclusion Criteria:

* age 60 years or more,
* residents of the study villages,
* no stroke,
* no significant disability,
* no dementia

Exclusion Criteria:

* age younger than 60 years,
* previous stroke,
* disabled,
* demented

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Social isolation and loneliness | one year
  The primary outcome is the change in social isolation and loneliness from baseline to 12 months. Social isolation will be measured using the Lubben Social Network Scale-6 (LSNS-6), which assesses the size and frequency of contact within family and friendship networks. Loneliness will be measured using the De Jong Gierveld Loneliness Scale, which evaluates emotional and social dimensions of perceived loneliness. Both instruments are validated for use in older adult populations. Scores will be collected at baseline, 6 months, and 12 months. The primary analysis will compare changes over time between the intervention community receiving the Social Connection Intervention Program (SCIP) and the comparison communities receiving usual activities.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar H Del Brutto, MD, Study Chair — Proyecto Atahualpa
Locations (1):
- Universidad Espiritu Santo, Samborondón, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No
participants names will be codified.

REFERENCES:
- [Result] Taylor HO, Cudjoe TKM, Bu F, Lim MH. The state of loneliness and social isolation research: current knowledge and future directions. BMC Public Health. 2023 Jun 1;23(1):1049. doi: 10.1186/s12889-023-15967-3. PMID 37264355